CLINICAL TRIAL: NCT05623943
Title: Comparison of Cerebral Artery Pressure Gradient and Cerebral Blood Flow Measured by Arterial Spin Labeling
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: National Key Research and Development Project, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: XWFFR-1
Record Dates: First submitted 2022-10-28; First posted 2022-11-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Ischemic; Intracranial Atherosclerosis
Keywords: Intracranial atherosclerotic diseases; Fractional Flow Reserve; intravascular pressure gradients; Cerebral blood flow; Arterial Spin Labeling
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICAS patients planning for endovascular treatment: Patients received pressure-wire-based intravascular pressure measurement and ASL measurement before and after operation.
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Patients treated with endovascular treatment, including balloon angioplasty alone and balloon angioplasty plus stenting.

SUMMARY:
The goal of this observational study is to explore the ability of intravascular pressure gradients to identify hemodynamic disturbance in patients with intracranial atherosclerotic diseases (ICAS). The main questions that aim to answer are:

* The correlation between intravascular pressure gradient and cerebral blood flow (CBF)
* The threshold for intravascular pressure gradients to predict hemodynamic disturbance in ICAS

Patients will undergo intravascular pressure measurement and arterial spin labeling (ASL) for CBF during pre- and post-operation respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40 years or older.
2. Patients with transient ischemic attack (TIA) or nondisabling ischemic stroke caused by a focal ICAS lesion located in intracranial anterior circulation (vertebral artery, basilar artery or intracranial internal carotid artery and their major branches).
3. 50% to 99% stenosis (calculated by modified WASID method) of responsible arterial occlusion, confirmed by digital subtraction angiography (DSA).
4. Informed of the study protocol and objectives.

Exclusion Criteria:

1. Non-atherosclerotic MCA stenosis
2. Combined with moderate or severe stenosis of other extracranial and intracranial arteries
3. Previous endovascular treatment or surgery for cerebrovascular diseases
4. Large cerebral infarction (more than 1/2 MCA perfusion area)
5. Combined with other neurological diseases, such as aneurysm, arteriovenous malformation, tumor, hydrocephalus, cerebral trauma, cerebral hemorrhage, multiple sclerosis, epilepsy and intracranial infection.
6. Vascular abnormality or stunting, resulting in the impossibility of endovascular intervention
7. Liver and kidney dysfunction, or severe allergy to the contrast agent
8. Severe coagulation dysfunction
9. Pregnancy or in the preparation for pregnancy
10. Patients who cannot tolerate or do not allow MR screening, including metal implanting and claustrophobia
11. Patients with severe dementia or mental disorders, who cannot cooperate with examination

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ICAS resorting to endovascular therapy in our center were recruited consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The relevance between intravascular pressure gradients and CBF | Post-operation, an average of 3 days
  Patients will be divided into 2 groups according to whether they have hemodynamic disorders before operation and improve after operation. Fractional flow reserve (FFR) measurement will be analyzed in each group.

SECONDARY OUTCOMES:
The difference of ASL-CBF between pre- and post-operation | Baseline and Post-operation, an average of 3 days
  The mean cerebral blood flow (CBF) of ipsilateral region of interest (ROI) in two different layers will be recorded as CBF in MCA perfusion area of this side. Relative CBF (rCBF) is defined as the ratio of the affected side CBF to the contralateral CBF. When preoperative rCBF<0.9 and postoperative rCBF≥0.9, the patient will be considered to have hemodynamic disorders and be improved post-operation.
The difference of FFR between pre- and post-operation | Baseline and Post-operation, an average of 3 days
  FFR measurement will be performed at rest by 0.014-inch pressure guide wires (C12008, Abbot St. Jude Medical, Minneapolis, MN, USA) designed for coronary diseases. The mean endovascular pressure of distal and proximal lesions will be measured and recorded as Pd and Pa, respectively. Pd/Pa and Pa-Pd will be calculated and recorded before and after endovascular treatment.
Any stroke or death in short term. | 30±5 days
Procedure-related complications | 30±5 days
  Any complications, related to manometry and treatment, will be recorded including arterial dissection, arterial perforation, acute vascular occlusion and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China